CLINICAL TRIAL: NCT05400213
Title: Randomized Controlled Trial of Wound Healing Following Tooth Extraction and Ridge Preservation Using Decalcified Freeze-dried Bone Allograft (DFDBA) Alone in Particulate Fiber Form and in Combination With Xenograft
Brief Title: Wound Healing Following Tooth Extraction and Ridge Preservation Using DFDBA Alone in Particulate Fiber Form and in Combination With Xenograft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20220346H
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Dental Extraction; Wound Heal
Keywords: Ridge preservation; Implant
MeSH Terms: interventions — Transplantation, Heterologous

STUDY DESIGN:
Intervention Model Description: 4 arm randomized controlled parallel study
Who Masked: Outcomes Assessor
Masking Description: Since the outcome of the study is the histologic healing, blinding of the surgeon is not necessary.
  Blinding is performed only for histomorphometric measurements. The person doing histomorphometric analysis is blinded as to study group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Group 1 Vallos (DCP) (Active Comparator): Subjects will be randomized into this group and receive DFDBA particulate alone
  Interventions: Device: Vallos (DCP)
- Group 2 Vallomix (DCF) (Active Comparator): Subjects will be randomized into this group and receive DFDBA fibers alone
  Interventions: Device: Vallomix (DCF)
- Group 3 Vallos-F (DPX) (Active Comparator): Subjects will be randomized into this group and receive Xenograft combined with DCP
  Interventions: Device: Vallos-F (DPX)
- Group 4 Vallomix-F (DFX) (Active Comparator): Subjects will be randomized into this group and receive Xenograft combined with DCF.
  Interventions: Device: Vallomix-F (DFX)

INTERVENTIONS:
Device: Vallos (DCP) — Demineralized freeze-dried bone allograft (DFBA) in a small particle form
  Other Names: DFDBA particulate
  Arms: Group 1 Vallos (DCP)
Device: Vallomix (DCF) — A combination of cow-derived xenograft and human-derived DFDBA particulate
  Other Names: Xenograft and human-derived DFDBA
  Arms: Group 2 Vallomix (DCF)
Device: Vallos-F (DPX) — Demineralized freeze-dried bone allograft (DFDBA) in a fiber form
  Other Names: DFDBA in fiber form
  Arms: Group 3 Vallos-F (DPX)
Device: Vallomix-F (DFX) — A combination of cow-derived xenograft and human-derived DFDBA fibers
  Other Names: Xenograft (Bio-Oss) combined with DFDBA fibers
  Arms: Group 4 Vallomix-F (DFX)

SUMMARY:
The primary aim of the study is to determine the amount of newly formed vital bone, residual graft material, and "connective tissue/other" 18 to 20 weeks after ridge preservation is performed using DFDBA fibers alone, DFDBA particulate alone, a combination of xenograft and DFDBA particulate, or a combination of xenograft and DFDBA fibers.

DETAILED DESCRIPTION:
The study plan is to extract non-molar teeth and graft with the various graft materials. Each subject will provide a single non-molar tooth site for study treatment. Following approx. 18-20 weeks of healing, the study team will harvest a core biopsy at the time of implant placement. The implant osteotomy is prepared with a trephine drill and the core inside the trephine is placed in 10% formalin for future processing and histomorphometric analysis. The core biopsy will be evaluated for the primary histologic outcome of % vital bone formation and the secondary histologic outcomes of % residual graft material, and % "CT/other" (fibrous tissue and marrow space). The study team will also evaluate the following secondary clinical outcomes using a custom measuring stent for each subject: change in ridge width; change in buccal ridge height and change in lingual ridge height. During the 18 to 20-week healing period, patients will be followed as needed per standard care to evaluate healing.

ELIGIBILITY:
Inclusion Criteria:

* One tooth, excluding molars, that has been identified by dental faculty as requiring a single tooth extraction
* A dental implant is indicated and treatment planned to replace the missing tooth
* Have adequate restorative space for a dental implant-retained restoration
* Have at least 10mm of alveolar bone height, without impinging on the maxillary sinus or inferior alveolar canal.
* Have a dehiscence of the buccal or lingual bony plate of the tooth socket extending no more than 50% of the total depth of the socket.
* Female patients who have undergone a hysterectomy, tubal ligation, or menopause, and non-pregnant women of child-bearing potential.
* Are nonsmokers or former smokers. Current smokers may be included if they smoke <10 cigarettes per day

Exclusion Criteria:

* Will not cooperate with the follow-up schedule.
* Patients will not be entered who are mentally incompetent, prisoners, or pregnant.
* Pregnant women or women intending to become pregnant during the study period (as confirmed verbally; an over the counter pregnancy test will be provided if pregnancy status is unknown or suspected).
* Patients who become pregnant during the study will be withdrawn and standard care will be delivered.
* Smokers who smoke >10 cigarettes per day
* Clinical and/or radiographic determinations which will preclude inclusion in this study are: Active infection other than periodontitis; Inadequate bone dimensions or restorative space for a dental implant; Presence of a disease entity, condition or therapeutic regimen which decreases probability of soft tissue and bony healing, e.g., poorly controlled diabetes, chemotherapeutic and immunosuppressive agents, autoimmune diseases, history of bisphosphonate use or long-term steroid therapy; Positive medical history of endocarditis following oral or dental surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Mealey, DDS, MS, Principal Investigator — University of Texas Health Science Center San Antonio; Angela Palaiologou-Gallis, DDS, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio (Dental School), San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared as summary results on ClinicalTrials.gov and in a peer-review journal.
Supporting Information: Study Protocol, SAP
Time Frame: After study completion and after data are analyzed.

REFERENCES:
- [Derived] Foster JE, Coleman CC, Palaiologou AA, Mealey BL. Healing following ridge preservation using demineralized allograft particles or fibers alone, and combined with xenograft. J Periodontol. 2025 Jul 24. doi: 10.1002/jper.11374. Online ahead of print. PMID 40702945

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients presented with one non-molar tooth that was indicated for extraction and planned for an implant restoration. Additional inclusion criteria included the following: 1) adequate restorative space for an implant restoration, 2) at least 10mm of alveolar ridge height before any vital structures, and 3) non-smokers or current smokers smoking <10 cigarettes per day.
Groups:
- Group 1 Vallos (DCP): Subjects will be randomized into one of the four groups and receive the corresponding material for ridge preservation following tooth extraction.
  Vallos: Demineralized freeze-dried bone allograft (DFBA) in a small particle form
- Group 2 Vallomix (DPX): Subjects will be randomized into one of the four groups and receive the corresponding material for ridge preservation following tooth extraction.
  Vallomix: A combination of cow-derived xenograft and human-derived DFDBA particulate
- Group 3 Vallos-F (DCF): Subjects will be randomized into one of the four groups and receive the corresponding material for ridge preservation following tooth extraction.
  Vallos-F: Demineralized freeze-dried bone allograft (DFDBA) in a fiber form
- Group 4 Vallomix-F (DFX): Subjects will be randomized into one of the four groups and receive the corresponding material for ridge preservation following tooth extraction.
  Vallomix-F: A combination of cow-derived xenograft and human-derived DFDBA fibers
Period: Overall Study
Arm/Group | Group 1 Vallos (DCP) | Group 2 Vallomix (DPX) | Group 3 Vallos-F (DCF) | Group 4 Vallomix-F (DFX)
Started | 24 | 27 | 24 | 27
Completed Histologic Analysis | 23 | 27 | 24 | 27
Completed Clinical Measurements | 24 | 26 | 23 | 26
Completed | 23 | 26 | 23 | 26
Not Completed | 1 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 Vallos (DCP) | Group 2 Vallomix (DPX) | Group 3 Vallos-F (DCF) | Group 4 Vallomix-F (DFX) | Total
Number analyzed (Participants) | 24 | 27 | 24 | 27 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (16.9) | 58.6 (16.8) | 55.9 (15.4) | 63.2 (9.6) | 60.17 (14.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 9 | 10 | 43
  Male | 9 | 18 | 15 | 17 | 59
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 24 | 27 | 24 | 27 | 102

OUTCOME MEASURES:

1. Primary Outcome: Percentage Vital Bone Formation
Description: Measure of percentage of vital bone formation from extraction to time of implant, this is a measure of how much bone has regenerated since the extraction to the surgery.
Time Frame: Wound healing time ( approximately 18 to 20 weeks)
Measure: Mean (Standard Deviation); unit: percentage of vital bone formation
Groups:
- Group 1 Vallos (DCP): Subjects will be randomized into this group and receive Vallos (DCP): Demineralized freeze-dried bone allograft (DFBA) in a small particle form
- Group 2 Vallos-F (DPX): Subjects will be randomized into this group and receive Vallos-F (DPX): Demineralized freeze-dried bone allograft (DFDBA) in a fiber form
- Group 3 Vallomix (DCF): Subjects will be randomized into this group and receive Vallomix (DCF): A combination of cow-derived xenograft and human-derived DFDBA particulate
- Group 4 Vallomix-F: Subjects will be randomized into this group and receive Vallomix-F (DFX): A combination of cow-derived xenograft and human-derived DFDBA fibers
Arm/Group | Group 1 Vallos (DCP) | Group 2 Vallos-F (DPX) | Group 3 Vallomix (DCF) | Group 4 Vallomix-F
Number analyzed (Participants) | 24 | 27 | 24 | 27
percentage of vital bone formation | 37.33 (14.31) | 40.76 (13.94) | 24.46 (13.75) | 23.85 (17.71)

2. Secondary Outcome: Percentage of Residual Graft Material
Description: Measure of percentage of residual graft material remaining at time of implant, this is the amount of graft material remaining from the original amount implanted during surgery.
Time Frame: Wound healing time ( approximately 18 to 20 weeks)
Measure: Mean (Standard Deviation); unit: percentage of residual graft material
Arm/Group | Group 1 Vallos (DCP) | Group 2 Vallos-F (DPX) | Group 3 Vallomix (DCF) | Group 4 Vallomix-F
Number analyzed (Participants) | 24 | 27 | 24 | 27
percentage of residual graft material | 16.25 (13.84) | 3.57 (2.78) | 23.39 (8.95) | 18.42 (10.24)

3. Secondary Outcome: Percentage of Connective Tissue at Time of Implant
Description: Measure of percentage of connective tissue (fibrous tissue and marrow space) at time of implant. This is the amount of connective tissue that is present at the time of surgery.
Time Frame: Baseline to 18-20 weeks
Measure: Mean (Standard Deviation); unit: percentage of connective tissue
Arm/Group | Group 1 Vallos (DCP) | Group 2 Vallos-F (DPX) | Group 3 Vallomix (DCF) | Group 4 Vallomix-F
Number analyzed (Participants) | 24 | 27 | 24 | 27
percentage of connective tissue | 46.41 (14.23) | 55.67 (14.28) | 52.03 (12.10) | 57.73 (14.72)

4. Secondary Outcome: Change in Ridge Width (Clinical Measurement)
Description: Measure of change in ridge width from extraction to healing time
Time Frame: Baseline to 18-20 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Group 1 Vallos (DCP) | Group 2 Vallos-F (DPX) | Group 3 Vallomix (DCF) | Group 4 Vallomix-F
Number analyzed (Participants) | 24 | 27 | 24 | 27
mm | -1.19 (0.94) | -1.02 (1.57) | -1.15 (1.02) | -1.00 (1.66)

5. Secondary Outcome: Change in Buccal Ridge Height (Clinical Measurement)
Description: Measure of change in buccal ridge height from extraction to healing time
Time Frame: Baseline to 18-20 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Group 1 Vallos (DCP) | Group 2 Vallos-F (DPX) | Group 3 Vallomix (DCF) | Group 4 Vallomix-F
Number analyzed (Participants) | 24 | 27 | 24 | 27
mm | -1.67 (1.99) | -0.85 (1.33) | -0.41 (2.19) | -1.08 (1.37)

6. Secondary Outcome: Change in Lingual Ridge Height (Clinical Measurement)
Description: Measure of change in lingual ridge height from extraction to healing time
Time Frame: Baseline to 18-20 weeks
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Group 1 Vallos (DCP) | Group 2 Vallos-F (DPX) | Group 3 Vallomix (DCF) | Group 4 Vallomix-F
Number analyzed (Participants) | 24 | 27 | 24 | 27
mm | -1.85 (1.63) | -0.75 (1.76) | -1.17 (1.72) | -1.75 (1.80)

ADVERSE EVENTS:
Time Frame: Baseline to 18-20 weeks
Groups:
- Group 1 Vallos: Subjects will be randomized into one of the four groups and receive the corresponding material for ridge preservation following tooth extraction.
  Vallos: Demineralized freeze-dried bone allograft (DFBA) in a small particle form
- Group 2 Vallos-F: Subjects will be randomized into one of the four groups and receive the corresponding material for ridge preservation following tooth extraction.
  Vallos-F: Demineralized freeze-dried bone allograft (DFDBA) in a fiber form
- Group 3 Vallomix: Subjects will be randomized into one of the four groups and receive the corresponding material for ridge preservation following tooth extraction.
  Vallomix: A combination of cow-derived xenograft and human-derived DFDBA particulate
- Group 4 Vallomix-F: Subjects will be randomized into one of the four groups and receive the corresponding material for ridge preservation following tooth extraction.
  Vallomix-F: A combination of cow-derived xenograft and human-derived DFDBA fibers
Arm/Group | Group 1 Vallos | Group 2 Vallos-F | Group 3 Vallomix | Group 4 Vallomix-F
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/27 | 0/24 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/27 | 0/24 | 0/27
Other Adverse Events (participants affected / at risk) | 0/24 | 0/27 | 0/24 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Vallos (N=24) | Group 2 Vallos-F (N=27) | Group 3 Vallomix (N=24) | Group 4 Vallomix-F (N=27)
Bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant experienced bleeding related to the dental procedure, rather than the intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT05400213/Prot_SAP_000.pdf